CLINICAL TRIAL: NCT01541397
Title: Bone Mineral Density in Adults With Hyperphenylalaninemia on Kuvan Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Heather Saavedra, Nutritionist; Department of Pediatrics Division of Genetics, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-11-0119
Record Dates: First submitted 2011-07-11; First posted 2012-03-01 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Hyperphenylalaninemia; Phenylketonuria
Keywords: Hyperphenylalaninemia; Phenylketonuria; Adults; Bone Mineral Density
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Kuvan treated (No Intervention): Adults with hyperphenylalaninemia who have are not receiving Kuvan therapy.
- Kuvan treated (Experimental): Adults with hyperphenylalaninemia who are treated with Kuvan (sapropterin).
  Interventions: Drug: Sapropterin

INTERVENTIONS:
Drug: Sapropterin — 20 mg/kg, orally, daily, 1 year or patient chooses to discontinue therapy
  Other Names: Kuvan
  Arms: Kuvan treated

SUMMARY:
Prospective study to compare the bone mineral density in adults with HPA on KUVAN™ therapy to those not on therapy. The investigators hypothesize that after one year of KUVAN™ therapy, there will be an improvement in their bone mineral density.

DETAILED DESCRIPTION:
Hyperphenylalaninemia (HPA) is a rare metabolic disorder caused by a deficiency of the enzyme phenylalanine hydroxylase (PAH) (NIH, October 16-18, 2000). Elevated plasma levels of phenylalanine (phe) cause mental retardation, microcephaly, delayed speech, seizures, eczema, and behavior abnormalities. Adequate control of the plasma levels of phe by a phe-restricted diet can prevent the developmental and behavioral problems.

The foundation of this diet is a phe-free metabolic medical product/formula made from free amino acids. Based on longitudinal studies, it has been reported that the most benefit is attained by individuals who maintain a phe-restricted diet throughout life. On December 13, 2007, KUVAN™ (sapropterin dihydrochloride) was approved by the FDA for the indication of reducing blood phe levels in patients with HPA due to BH4 responsive PKU, in conjunction with a phe restricted diet (BioMarin Pharmaceutical Inc., Investigator's Brochure March 25, 2008). Studies were performed to determine a definition of response to KUVAN™. In a phase 2 clinical trial in 2007, Burton, et. al. defined a Kuvan™ responder as having a 30% or greater improvement in blood phenylalanine levels compared to baseline after 8 days of drug therapy.

Kuvan™ has been shown to improve phenylalanine tolerance in some individuals with HPA. This drug enables these individuals to consume more protein from natural sources. However, there have been no research studies assessing the effects of KUVAN™ along with liberalization of the diet on bone mineral density.

The investigators propose a prospective study to compare the bone mineral density in adults with HPA on KUVAN™ therapy to those not on therapy. The investigators hypothesize that after one year of KUVAN™ therapy, there will be an improvement in their bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hyperphenylalaninemia at birth
* Age between 18 and 50 years
* Participated in study HSC-MS-110-0262

Exclusion Criteria:

* Peri-menopausal and menopausal women will be excluded because this is a time of increased bone loss related to hormonal mediated factors.
* Patients taking bisphosphonates because it alters bone density. Therefore, bone mineral density would reflect the biphosphonate intervention rather than their true status.
* Pregnant women due to the hazard of radiation exposure during a DXA scan. In addition women who have been pregnant or who have breastfed within one year of study enrollment will be excluded because these are periods of rapid bone loss which would not reflect the entity under study but would serve to confound the data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather W Saavedra, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Kuvan Treated | Kuvan Treated
Started | 4 | 2
Completed | 0 | 0
Not Completed | 4 | 2
Not completed — Study ended prior to data collection | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Kuvan Treated | Kuvan Treated | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: A DXA scan will be conducted one year after Kuvan therapy is initiated.
Time Frame: 1 year after initiation of Kuvan therapy
Population: Zero participants were analyzed because the study was ended early (due to an insufficient number of enrolled participants).
Arm/Group | Non-Kuvan Treated | Kuvan Treated
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Plasma Amino Acid Profile
Description: Evaluation of levels of plasma amino acids.
Time Frame: every three months up to 1 year
Population: as for outcome 1
Arm/Group | Non-Kuvan Treated | Kuvan Treated
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Diet Analysis
Description: Subjects will provide a 3 day diet record for every plasma amino acid evaluation. Diets will be analyzed to determine phenylalanine, protein, calories, fat, vitamins and minerals.
Time Frame: every 3 months up to 1 year
Population: as for outcome 1
Arm/Group | Non-Kuvan Treated | Kuvan Treated
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Plasma Phenylalanine Levels
Description: Plasma phenylalanine levels will be monitored to determine effectiveness of Kuvan therapy.
Time Frame: weekly for 6 weeks, then at least every three months up to 1 year
Population: as for outcome 1
Arm/Group | Non-Kuvan Treated | Kuvan Treated
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Non-Kuvan Treated | Kuvan Treated
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes